CLINICAL TRIAL: NCT03993951
Title: The Use of Information and Communications Technology in Family Service Agencies
Brief Title: Information and Communications Technology in Family Services
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UW18-073
Record Dates: First submitted 2018-07-16; First posted 2019-06-21 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Family Research
Keywords: Family

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ICT System — Update the Information and Communications Technology System in Family Service Agencies

SUMMARY:
In the past few decades, Information and Communications Technology (ICT) have rapidly developed as effective, and probably the most cost-effective, tools to connect most, if not all, aspects of family lives.

To promote family harmony, The Hong Kong Jockey Club Charities Trust has initiated the Jockey Club SMART Family-Link Project in collaboration with The University of Hong Kong (HKU) and NGOs. This project, making effective use of information and communications technology (ICT) and data analytics, is aimed at helping 26 NGO-operated Integrated Family Service Centres and Integrated Service Centres (Centres) enhance the quality and efficiency of their family service. The project is also aimed at building the capabilities of front-line workers so as to achieve the goal of enhancing family well-being.

This study aim to gain a deeper and more comprehensive understanding of the current level of ICT use by the providers of family services in Hong Kong, and their anticipated future direction regarding ICT use. In-depth and focus group interviews are conducted for the stakeholders (such as heads of service, programme directors, counsellors and service users) from the non-government organisations (NGOs) and the Social Welfare Department. The interviews help identify the concerns of social service and related workers and the needs of the participating NGOs in the development of the ICT system and the application in their services. The needs and concerns of the stakeholders in using ICTs in family services will be identified. It can facilitate the planning and designing of the system, the community programmes, and the training and sharing platform. The system will better fit the needs of the social service sector. In addition, the impact of JC SMART Family-Link Project on the stakeholder in family services will be evaluated through questionnaire survey and focus group interviews.

DETAILED DESCRIPTION:
Information and Communications Technologies (ICTs) as a global trend refers to a cluster of technologies that are used to share, distribute, gather, and communicate information. ICTs encompass hardware that is often Internet capable such as computers, smart phones, and tablets, as well as the software and applications, such as email, social media sites, and video conferencing that are used on these devices. In Hong Kong, as of March 2016, the number of mobile service subscribers was 16.72 million, representing one of highest penetration rates in the world at about 228.3 per cent; amongst these subscribers, 14.69 million were 3G/ 4G service customers. As of March 2016, a surge to 20,557 Terabytes (or an average of 1,358 Megabytes per 2.5G/3G/4G mobile user) was recorded for local mobile data usage, representing a growth of 1.18 times and 1.58 times over the same period in 2015 and 2014 respectively.

In light of the review on family services in Hong Kong in 2000, pilot projects on the Integrated Family Service Centre (IFSC) service mode, were conducted in 2002. The Review report "Building Effective Family Services: Review on the Implementation of the IFSC Service Mode" stated that the IFSC service mode is an appropriate service mode for public-funded family services in Hong Kong. However, the Review also identified factors hindering the delivery of IFSC services. These hindering factors are the namely poor accessibility of some IFSCs, heavy workload, and stigmatisation. With the use of ICT, these hindering factors can be overcome, thus improving the IFSC service mode. The Review also recommended that "IFSCs should explore service enhancement through appropriate use and sharing of information technology."

To gain a more comprehensive understanding of the current level of ICT use by providers of family services in Hong Kong, and their anticipated future direction regarding ICT use, focus group interviews are conducted with various stakeholders, including heads of service and programme directors at Hong Kong NGOs running IFSCs, and social service workers and service users of various IFSCs. Focus group interviews and survey questionnaires for service providers and service users are used to collect the information on the view and use of ICT in their daily practice.

The Hong Kong Jockey Club Charities Trust has initiated the Jockey Club SMART Family-Link Project in collaboration with The University of Hong Kong (HKU) and NGOs to promote the effective use of information and communications technology (ICT) and data analytics in family services. This project is aimed at helping 26 NGO-operated Integrated Family Service Centres and Integrated Service Centres (Centres) devise an innovative and evidence-based family service delivery model that leverages the effective use of ICT and data analytics and enhance the quality and efficiency of their family service.

This study aims to (i) understand the current practice of ICT use in family services and identify the needs and concerns of the stakeholders (heads of service, programme directors, counsellors, social service and related workers, and service users) on using ICTs in family services; and (ii) assess the impact of the Jockey Club SMART Family-Link Project.

ELIGIBILITY:
Inclusion Criteria:

* Stakeholders from the social service sector.
* Aged 18 years or older
* Cantonese speaking

Exclusion Criteria:

- Subjects who fail to meet the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Social and service-related workers including heads of service, programme directors, counsellors and service users
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in views of ICTs use in family services from baseline at 1 year | baseline and year 1
  Outcome based questions will be used to assess the views of social and service-related workers on using ICTs in family services. Question scores for range from 0 to 10. The higher score indicates the better outcome performance
The change in behaviours of using ICTs in family services from baseline at 1 year | baseline and year 1
  Outcome based questions will be used to assess the behaviours of social and service-related workers on using ICT in family services. Question scores range from 0 to 10. The higher score indicates the better outcome performance

SECONDARY OUTCOMES:
The views of ICTs use in family services | year 2 and year 3
  Outcome based questions will be used to assess the views of social and service-related workers on using ICTs in family services. Question scores for range from 0 to 10. The higher score indicates the better outcome performance
The behaviours of using ICT in family services | year 2 and year 3
  Outcome based questions will be used to assess the behaviours of social and service-related workers on using ICTs in family services. Question scores for range from 0 to 10. The higher score indicates the better outcome performance
The knowledge of using ICT in family services | baseline, year 1, year 2 and year 3
  Outcome based questions will be used to assess the knowledge of social and service-related workers on using ICT in family services. Question scores range from 0 to 10. The higher score indicates the better outcome performance
The attitude of using ICT in family services | baseline, year 1, year 2 and year 3
  Outcome based questions will be used to assess the attitude of social and service-related workers on using ICT in family services. Question scores range from 0 to 10. The higher score indicates the better outcome performance
The perceived effects in related to using ICT in family services | baseline, year 1, year 2 and year 3
  Outcome based questions will be used to assess the perceived effects on using ICT in family services. Question scores range from 0 to 10. The higher score indicates the better outcome performance

CONTACTS AND LOCATIONS:
Overall Officials: Tai-hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Social service sector, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sit SMM, Lai AYK, Kwok TO, Wong HW, Wong YL, Lam EYW, Chan JYW, Kong FSW, Cham K, Ng CKK, Yip T, Tsui TSY, Wong CM, Wong BCL, Tang WY, Yam PW, Chui M, Wan A, Kwok YK, Lam TH. Process Evaluation and Experience Sharing on Utilizing Information Communication Technologies and Digital Games in a Large Community Family Health Event: Hong Kong Jockey Club SMART Family-Link Project. Front Public Health. 2020 Dec 22;8:579773. doi: 10.3389/fpubh.2020.579773. eCollection 2020. PMID 33415096
- See also: Description: The World Bank, 2016. Internet users (per 100 people). — http://data.worldbank.org/indicator/IT.NET.USER.P2?end=2014&start=1990